CLINICAL TRIAL: NCT05346510
Title: Evaluation of Axillary Lymph Nodes Using Prone Positioning Computed Tomography Scan and Ultrasound in Patients With Breast Cancer
Brief Title: Prone Positioning CT Scan and Ultrasound Assessing Axillary Lymph Nodes in Patients With Breast Cancer Official Title: Evaluation of Axillary Lymph Nodes Using Prone Positioning Computed Tomography Scan and Ultrasound in Patients With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Jianyi Li, Principal Investigator, Shengjing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Shengjing-LJY07
Record Dates: First submitted 2022-04-19; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; axillary lymph node; prone positioning computed tomography; ultrasound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ALND Group (Experimental): ALND is performed in patients with positive axillary lymph nodes on CT scan and on AAUS.
  Interventions: Procedure: ALND Group
- pALND Group (Experimental): pALND is performed in patients with negative axillary lymph nodes on CT scan but positive on AAUS.
  Interventions: Procedure: ALND Group
- SLNB Group (Experimental): SLNB will be performed for those with negative axillary lymph nodes on CT scan and on AAUS.
  Interventions: Procedure: ALND Group

INTERVENTIONS:
Procedure: ALND Group — ALND is performed in patients with positive axillary lymph nodes on CT scan and on AAUS. pALND is performed in patients with negative axillary lymph nodes on CT scan but positive on AAUS.SLNB will be performed for those with negative axillary lymph nodes on CT scan and on AAUS.
  Other Names: pALND Group; SLNB Group

SUMMARY:
The early diagnosis and evaluation of breast cancer is of great significance to its treatment and prognosis. Among the multiple factors affecting the prognosis, the degree of axillary lymph node metastasis is one of the most vital factors.

Accurately understanding the status of axillary lymph nodes prior to surgery allows better prediction of staging, enables correct treatment plans, and guides the scope of node dissection during surgery. For patients with early breast cancer or clinically negative axillary lymph nodes, sentinel lymph node biopsy (SLNB) can largely avoid complications such as upper extremity lymphedema caused by axillary lymph node dissection (ALND). Thus, clinical identification of negative lymph nodes becomes more valuable. Based on clinical verification, the NCCN guidelines (edition 2019) made the following recommendation: SLNB is performed for patients with clinically negative axillary lymph nodes, and the biopsy findings determine whether ALND is included; ALND is performed for patients with clinically positive axillary nodes. Currently, imaging examinations have limitations is assessing axillary lymph nodes. Finding an accurate and non-invasive method in preoperative axillary assessment has been a project that needs to be urgently addressed. Ultrasonography has advantages in its simplicity, non-invasiveness, economy, and on radiation, however it is highly subjective, dependent upon examiner's experience and knowledge, and is difficult to detect deeper and small lesions. Molybdenum Target examination plays an important role in diagnosis of breast cancer, however it is expensive and limited in evaluating the whole axilla. PET-CT is restricted by its high cost and is not a routine examination in China.

Therefore, computed tomography (CT) scan is more advantageous in determination of lymph node metastasis. The 2014 GORO KUTOMI study suggested that lymph node morphology assessed as clear by preoperative CT was an independent predictor of sentinel lymph node metastasis. CT scan can not only evaluate the presence or absence of distant metastasis and pectoralis muscle invasion, but also provide intuitive, accurate and detailed evaluation of axillary, supraclavicular, and pectoralis major intramuscular lymph nodes. The diagnostic criteria of magnetic resonance imaging (MRI) is relatively vague; CT can also obtain imaging data of the lungs, mediastinum, whereas MRI has no such function. Based on previous studies, we will further explore and evaluate axillary node status using prone positioning CT scan and ultrasound in patients with breast cancer.

DETAILED DESCRIPTION:
A total of 500 patients who are newly diagnosed with operable breast cancer in Liaoning Oncology Hospital are approached and recruited. Inclusion criteria: 1. preoperative chest CT and axillary Doppler ultrasound examination in the prone position; 2. perform ALND; 3. regular follow-up post surgery, short-term and long-term. Exclusion criteria: history of other benign or malignant tumors causing axillary lymphadenopathy.

Comparisons are made:

A: between suspiciously positive and suspiciously negative axillary lymph nodes B: between LNSD positive among suspiciously positive axillary lymph nodes and negative axillary lymph nodes f C: between positive and negative AAUS D: between positive and negative AAUS among negative lymph nodes detected by CT scan E: between positive and negative AAUS among lymph nodes with negative LNSD

Chi-square test and t test are used to assess statistical significance between groups.

Methods: Lymph node short diameter (LNSD) is measured using CT scan imaging (LNSD > 1cm is considered positive), axillary lymph node status is assessed according to axillary lymph node Doppler ultrasound. ALND will be performed in patients with positive axillary lymph nodes on CT scan; PALND will be performed for those with negative axillary lymph nodes on CT scan but positive on AAUS; SLNB will be performed for those with negative axillary lymph nodes on CT scan and on AAUS.

The prognosis in each patient group is to be evaluated by short-term observational indicators (e.g. lymphedema and/or status of axillary lymphatic return), and long-term indicators (e.g. lymphedema and/or axillary lymph node recurrence). The accuracy of CT scan assessing positive lymph nodes and positive AAUS will be evaluated according to the postoperative histology results.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative chest CT and axillary Doppler ultrasound examination in the prone position
* Perform ALND
* Regular post surgery follow-up (short-term and long-term)

Exclusion Criteria:

•History of other benign or malignant tumors causing axillary lymphadenopathy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Agreement rates with postoperative histology | Two weeks
  The accuracy of CT scan detecting positive axillary lymph node and positive AAUS is assessed by the postoperative histology results

SECONDARY OUTCOMES:
The incidence of postoperative lymphedema (short-term observational indicator) | Two years
  The purpose of SLNB is to reduce the scope of axillary lymph node dissection, therefore reduce the occurrence of complications.
Axillary recurrence rate | Five years
  Axillary recurrence rate as a long-term observational indicator

CONTACTS AND LOCATIONS:
Overall Officials: Jianyi Li, Dr, Principal Investigator — Cancer Hospital of China Medical University, Liaoning Cancer Hospital
Locations (1):
- Liaoning Oncology Hospital, Shenyang, Liaoning, China